CLINICAL TRIAL: NCT02514460
Title: Clinical Study of Stent Versus Direct Atherectomy to Treat Lower Limb Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z141107002514063
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2015-12

CONDITIONS: Atherosclerosis; Ischemia
Keywords: stents; atherectomy; femoral artery; popliteal artery
MeSH Terms: conditions — Atherosclerosis; Ischemia | interventions — Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: Stents (Active Comparator): Stents group
  Interventions: Device: Stent
- Intervention: Atherectomy (Active Comparator): Direct Atherectomy group
  Interventions: Device: plaque excision system

INTERVENTIONS:
Device: plaque excision system
  Arms: Intervention: Atherectomy
Device: Stent
  Arms: Intervention: Stents

SUMMARY:
This is a randomized study comparing stent and plaque excision systems in treatment of lower limb (superficial femoral or popliteal artery) ischemia.

DETAILED DESCRIPTION:
This is a randomized study comparing stent and plaque excision systems in treatment of diabetic lower limb (superficial femoral or popliteal artery) ischemia.

ELIGIBILITY:
Inclusion Criteria:

Provides written informed consent Willing to comply with follow-up evaluations at specified times Has claudication or rest pain due to peripheral arterial disease Disease located within the femoropopliteal artery Patient has a de novo or restenotic lesion(s) with >50% stenosis documented angiographically and no prior stent in the target lesion.

Patient has symptoms of peripheral arterial disease classified as Rutherford Category 2 or greater.

Exclusion Criteria:

Previously implanted stent(s) or stent graft(s) in target leg Life expectancy less than 12 months Has any planned surgical or endovascular intervention of target vessel 30 days before or after index procedure Thrombophlebitis, uremia, or deep venous thrombus, within past 30 days. Receiving dialysis or immunosuppressant therapy. Recent stroke within past 90 days. Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix®) or ticlopidine (Ticlid®), heparin, Nitinol (nickel titanium), contrast agent, that cannot be medically managed.

Tissue loss due to ischemic disease (Rutherford/Becker category 5 or 6) Serum creatinine level >/= 2.5 mg/dl at time of screening visit Known or suspected active infection at the time of the procedure Bleeding diathesis Patient is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol.

Patient is known to be pregnant, incarcerated, mentally incompetent, and/or alcohol or drug abuser.

Patient is currently participating in any other investigational drug or medical device study that has not completed primary endpoint(s) evaluation or clinically interferes with the endpoints from this study or future participation in such studies prior to the completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
12-month Primary Patency Rate | 12 months
  Primary patency is defined as no significant reduction of flow detectable by Duplex ultrasound through the index lesion and no further clinically driven target vessel revascularization performed in the interim. Significant reduction of flow is binary restenosis defined as the diameter stenosis >50% with a peak systolic velocity ratio >2.4 as measured by Duplex ultrasound.
12-month Limb Salvage Rate | 12 months
  Limb Salvage is defined as the freedom from secondary major amputation

SECONDARY OUTCOMES:
Index Limb Ischemia at 6-month Follow up | 6 months
  Index Limb Ischemia is defined by Rutherford/Becker Classification categories 3 through 6.
Index Limb Ischemia at 12-month Follow up | 12 months
  Index Limb Ischemia is defined by Rutherford/Becker Classification categories 3 through 6.
Major Adverse Events at 12-month Post Procedure | 12 months
  Major adverse events included death, index limb ischemia, index limb amputation, clinically driven target lesion revascularization , and significant embolic events, which were defined as causing end-organ damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Gu Yong Quan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yongquan G, Lianrui G, Lixing Q, Xuefeng L, Zhu T, Shijun C, Yingfeng W, Jianming G, Jian Z, Zhonggao W. Plaque excision in the management of lower-limb ischemia of atherosclerosis and in-stent restenosis with the SilverHawk atherectomy catheter. Int Angiol. 2013 Aug;32(4):362-7. PMID 23822938